CLINICAL TRIAL: NCT03948698
Title: Evaluation of the Catalyzing Pediatric TB Innovations Project: A Pre- and Post-Implementation Assessment Across Ten Countries
Brief Title: TB Innovation Project: A Pre- and Post- Implementation Assessment (TIPPI)
Acronym: TIPPI
Status: Completed | Type: Observational
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: EG0209
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Results first posted 2021-12-20 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Tuberculosis; Pediatric
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Innovative approached to pediatric TB care — Includes integration of TB care in non-TB entry points in facilities, decentralization from higher level clinics to lower levels, strengthening screening activities and building diagnosis and treatment capacity among healthcare workers
  Other Names: Integration and decentralization

SUMMARY:
This evaluation will be conducted in ten countries involved in the Catalyzing Pediatric TB Innovation (CaP-TB) project: Cameroon, Cote D'Ivoire, Democratic Republic of Congo, Kenya, Lesotho, Malawi, Tanzania, Uganda, Zimbabwe and India. The CaP-TB project is a project designed to use innovative methods and capacity building to strengthen the health systems of developing countries in terms of pediatric TB case detection, early accurate diagnosis and effective treatment. This project is funded by Unitaid and is implemented by Elizabeth Glaser Pediatric AIDS Foundation.

EGPAF proposes to evaluate the implementation of CaP-TB in up to 450 sites in ten participating countries. This evaluation will assess the effects of CaP-TB innovative interventions on selected service delivery outcomes as compared to routine TB program in a sub-set of project sites in the ten countries.

DETAILED DESCRIPTION:
This pre-post quasi-experimental evaluation study will be conducted in ten countries involved in the Catalyzing Pediatric TB Innovation (CaP-TB) project: Cameroon, Cote D'Ivoire, Democratic Republic of Congo, Kenya, Lesotho, Malawi, Tanzania, Uganda, Zimbabwe and India. The CaP-TB project is a project designed to use innovative methods and capacity building to strengthen the health systems of developing countries in terms of pediatric TB case detection, early accurate diagnosis and effective treatment. This project is funded by Unitaid headquartered in Geneva, Switzerland and is implemented by Elizabeth Glaser Pediatric AIDS Foundation (EGPAF) with headquarters in Washington, D.C. and Geneva and 10 country offices. This study will assess the effects of CaP-TB innovative interventions on selected service delivery outcomes as compared to routine TB program in a sub-set of project sites in ten countries.

The CaP TB project is a 4-year (October 1, 2017-September 30, 2021) Unitaid-funded project to improve pediatric TB outcomes by introducing integrated and decentralized models of pediatric TB care and strengthening access to WHO-recommended drugs and diagnostics. Integration refers to supporting TB activities, such as screening and TB sample collection for children, into non-TB health care services, such as general pediatric outpatient clinics. Decentralization refers to moving pediatric TB services from higher levels of health clinics to lower levels.

Objectives of the study

To evaluate the CaP TB project on the below TB service indicators and clinical outcomes for children 0-14 in facilities implementing the CaP TB project:

* Number and proportion of children screened for TB among clinic attendees
* Number and proportion of presumptive TB cases referred for lab-based TB diagnosis
* Number and proportion of pediatric presumptive TB cases who are tested with Xpert
* Number and proportion (out of all children screened) of pediatric cases diagnosed with active TB disease
* Time between when a child is identified as a presumptive TB case and when the child is diagnosed with TB
* Number and proportion of pediatric TB cases started on DS-TB treatment
* Time between when a child is identified as a presumptive TB case and when the child is initiated on TB treatment
* Number and proportion of pediatric DS-TB cases or cases treated with first-line TB treatment who achieve treatment success
* Number and proportion of all TB index cases for whom successful contact tracing has been done
* Number and proportion of pediatric household contacts who are negative to TB screening

Study data

Pre-intervention retrospective data collection

Under the standard of care condition (baseline), the investigators will:

* Capture data that will answer the TB service indicators and clinical outcomes listed in the primary objectives.
* Capture key data points that will be needed to estimate project targets In each site, trained data collectors will retrospectively extract data from appropriate registers, logs, and in some cases patient files, for a period of 12 months starting 6 months before the start date of data extraction.

After the implementation of the CaP TB project, prospective data will be collected by project-specific data collection tools and/or from existing registers. Whenever possible, the CaP TB data collection will use existing site level data collection tools to gather the data for the project.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric TB patients (0-14 years of age) in CaP TB project sites in any of the 10 countries and receive TB screening (including screening, diagnosis and treatment for active TB, and provision of TB preventive therapy).
* All pediatric TB patients (0-14 years of age) in CaP TB project sites in any of the 10 countries and receive TB diagnosis
* All pediatric TB patients (0-14 years of age) in CaP TB project sites in any of the 10 countries and receive TB treatment for active TB
* All pediatric TB patients (0-14 years of age) in CaP TB project sites in any of the 10 countries and receive TB preventive therapy

Exclusion Criteria:

• All pediatric TB patients who enter CaP TB project site in any of the 10 countries and who are above 15 years old

Max Age: 14 Years | Sex: All
Age Groups: Child
Study Population: All pediatric TB patients (0-14 years of age) who present to a CaP TB project site in any of the 10 countries and receive TB services (including screening, diagnosis and treatment for active TB, and provision of TB preventive therapy).
Sampling Method: Non-Probability Sample
Enrollment: 4159533 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Cohn, MD, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation; Martina Casenghi, PhD, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation
Locations (10):
- Sites in Centre, Littoral and West regions, Djoungolo, Cameroon
- Adjame-Plateau-Attecoube, Abobo Est,Anyama , Koumassi-Port Bouet-Vridi, Treichville-Marcory, Abidjan, Côte d’Ivoire
- Bandalungwa,Binza Meteo,Kikimi,Kingasani,Kinshasa, Lingwala, Masina II, Mont Ngafula II, Ndjili, Kinshasa, Democratic Republic of the Congo
- Sites in Maharashtra State, Telangana State, Andhra Pradesh, Hyderabad, India
- Turkana County and Homabay County sites, Nairobi, Kenya
- Berea, Maseru, Mageteng, Leribe, Mohale's Hoek sites, Maseru, Lesotho
- Central Region, Southern region sites, Dedza, Malawi
- Singida, Tabora sites, Singida, Tanzania
- Mbarara sites, Mbarara, Uganda
- Harare, Manicaland, Matabeleland South, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lemaire JF, Cohn J, Kakayeva S, Tchounga B, Ekouevi PF, Ilunga VK, Ochieng Yara D, Lanje S, Bhamu Y, Haule L, Namubiru M, Nyamundaya T, Berset M, de Souza M, Machekano R, Casenghi M; CaP-TB Study team. Improving TB detection among children in routine clinical care through intensified case finding in facility-based child health entry points and decentralized management: A before-and-after study in Nine Sub-Saharan African Countries. PLOS Glob Public Health. 2024 Feb 5;4(2):e0002865. doi: 10.1371/journal.pgph.0002865. eCollection 2024. PMID 38315700
- [Derived] Mafirakureva N, Mukherjee S, de Souza M, Kelly-Cirino C, Songane MJP, Cohn J, Lemaire JF, Casenghi M, Dodd PJ. Cost-effectiveness analysis of interventions to improve diagnosis and preventive therapy for paediatric tuberculosis in 9 sub-Saharan African countries: A modelling study. PLoS Med. 2023 Sep 6;20(9):e1004285. doi: 10.1371/journal.pmed.1004285. eCollection 2023 Sep. PMID 37672524

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study does not have a set number of participants. The number of participants is number of children screened.
Groups:
- CaP TB TIPPI Study: No new information to report
Period: Overall Study
Arm/Group | CaP TB TIPPI Study
Started | 4749072
Completed | 4749072
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | CaP TB TIPPI Study
Number analyzed (Participants) | 2318
Age, Categorical [Count of Participants; unit: Participants] — Please note that the baseline data for this study was collected retrospectively using existing registers in health facilities, so the design does not compare the same exact children pre-post intervention. The baseline values that are entered here is what was available in countries at the time of the baseline data collection and these numbers will be different with the intervention data that is entered in other sections.
  Participants
    <=18 years | 2318
    Between 18 and 65 years | 0
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1163
  Male | 1155
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Cameroon | 159
  Malawi | 167
  Côte D'Ivoire | 247
  Congo, The Democratic Republic of the | 709
  Tanzania | 335
  Uganda | 92
  Zimbabwe | 281
  Kenya | 212
  Lesotho | 116

OUTCOME MEASURES:

1. Primary Outcome: Children Screened for TB
Description: Number and proportion of children (age 0-14) screened for TB among clinic attendees
Time Frame: December 2018-September 2021
Population: The number of participants analyzed, 7198865, is the clinic attendees and 4749072 is number of children screened. 4749072 is the number indicated in the participant flow because this data is generated by the study. Clinic attendees data is already available in health facilities.
Measure: Count of Participants; unit: Participants
Arm/Group | CaP TB TIPPI Study
Number analyzed (Participants) | 7198865
Participants | 4749072

2. Primary Outcome: Children With Presumptive TB
Description: Among those screened the number and proportion of children presumed to have TB.
Time Frame: December 2018-September 2021
Population: The number Started in the participant flow was revised and both values are equal
Measure: Count of Participants; unit: Participants
Arm/Group | CaP TB TIPPI Study
Number analyzed (Participants) | 4749072
Participants | 60250

3. Primary Outcome: Children With Presumptive TB Referred for Lab-based TB Diagnosis
Description: Number and proportion of presumptive TB cases referred for lab-based TB diagnosis
Time Frame: December 2018-September 2021
Measure: Count of Participants; unit: Participants
Arm/Group | CaP TB TIPPI Study
Number analyzed (Participants) | 60250
Participants | 49022

4. Primary Outcome: Children With Presumptive TB Tested Using GeneXpert
Description: Number and proportion of pediatric (0-14 years) presumptive TB cases who are tested with GeneXpert
Time Frame: December 2018-September 2021
Measure: Count of Participants; unit: Participants
Arm/Group | CaP TB TIPPI Study
Number analyzed (Participants) | 60250
Participants | 35554

5. Primary Outcome: Children Initiated on TB Preventive Therapy
Description: Number and proportion of pediatric patients started on preventive therapy of those who are eligible for preventive therapy
Time Frame: December 2018-September 2021
Measure: Count of Participants; unit: Participants
Arm/Group | CaP TB TIPPI Study
Number analyzed (Participants) | 36026
Participants | 28762

6. Primary Outcome: Children Completing TB Preventive Therapy
Description: Number and proportion of pediatric patients on preventive treatment who completed therapy
Time Frame: December 2018-September 2021
Population: Please note the number this measure is different than the one indicated for Children Initiation on PT because here we report Children that were initiated on PT with expected outcomes (i.e. 6 months of preventive therapy)
Measure: Count of Participants; unit: Participants
Arm/Group | CaP TB TIPPI Study
Number analyzed (Participants) | 28762
Participants | 22590

7. Primary Outcome: Children Diagnosed With Active TB
Description: Number of pediatric cases diagnosed with active TB disease among children with presumptive TB
Time Frame: December 2018-September 2021
Measure: Count of Participants; unit: Participants
Arm/Group | CaP TB TIPPI Study
Number analyzed (Participants) | 60250
Participants | 11078

8. Primary Outcome: Children Initiated on TB Treatment
Description: Number and proportion of pediatric TB cases started on DS-TB treatment
Time Frame: December 2018-September 2021
Measure: Count of Participants; unit: Participants
Arm/Group | CaP TB TIPPI Study
Number analyzed (Participants) | 11078
Participants | 10834

9. Primary Outcome: Children Achieving Treatment Success
Description: Number and proportion of pediatric DS-TB cases who achieve treatment success
Time Frame: December 2018-September 2021
Population: Please note that this measure if different than the one reported in Children initiated in DS TB treatment because this number only includes children with expected treatment outcomes (i.e completing 6 months treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | CaP TB TIPPI Study
Number analyzed (Participants) | 7221
Participants | 6553

10. Primary Outcome: TB Contacts Successfully Traced
Description: Number and proportion of all TB index cases for whom successful contact tracing has been done
Time Frame: December 2018-September 2021
Measure: Count of Participants; unit: Participants
Arm/Group | CaP TB TIPPI Study
Number analyzed (Participants) | 63314
Participants | 20998

11. Primary Outcome: TB Contacts Screened Negative for TB
Description: Number and proportion of pediatric household contacts who are negative to TB screening
Time Frame: December 2018-September 2021
Population: The overall number of participants analyzed here would be the number of contacts screened.
Measure: Count of Participants; unit: Participants
Arm/Group | CaP TB TIPPI Study
Number analyzed (Participants) | 48907
Participants | 37774

12. Primary Outcome: TB Contacts Eligible for Preventive Therapy
Description: Number and proportion of screened negative pediatric contacts eligible for preventive therapy
Time Frame: December 2018-September 2021
Population: Please note that these numbers will differ from the numbers reported on previous measures related to preventive therapy because these numbers only include contact tracing whereas previously reported measures included both TB contacts and people coming from HIV clinics
Measure: Count of Participants; unit: Participants
Arm/Group | CaP TB TIPPI Study
Number analyzed (Participants) | 37774
Participants | 19630

ADVERSE EVENTS:
Description: Please note that that this study does not monitor for adverse events because it does not introduce new treatment, etc. It is introducing a more intensified screening for TB and then monitors routine clinical screening procedures.
Groups:
- CaP TB TIPPI Study: No arms to report
Arm/Group | CaP TB TIPPI Study
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/98/NCT03948698/Prot_SAP_000.pdf